CLINICAL TRIAL: NCT03781700
Title: The Facial Nerve Palsy And Cortisone Evaluation (FACE) Study in Children: A Randomized Double-blind, Placebo-controlled, Multicenter Trial
Brief Title: Evaluation of Cortisone Treatment in Children With Acute Facial Nerve Palsy
Acronym: FACE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Barbro Hedin Skogman, MD, Assistant Professor, Dalarna County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FACE-01; 2017-004187-35 (EudraCT Number)
Record Dates: First submitted 2018-12-14; First posted 2018-12-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Facial Palsy; Facial Nerve Diseases; Borrelia Infection of Central Nervous System; Bell Palsy
Keywords: Children; Paediatric
MeSH Terms: conditions — Facial Paralysis; Facial Nerve Diseases; Bell Palsy | interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone (Experimental): Prednisolone
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Placebo oral tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Prednisolone — Prednisolone 5 milligram tablets, 1 milligram per kilogram bodyweight per orally per day during 10 days, maximum 50 milligram per day.
  Other Names: Batch 18A71, Orifarm Generics A/S
  Arms: Prednisolone
Drug: Placebo Oral Tablet — Placebo tablets with identical appearance to the experimental drug
  Other Names: Batch 18A61, Orifarm Generics A/S
  Arms: Placebo

SUMMARY:
Acute facial nerve palsy occur in 10-20/100 000 children/year in Sweden. About 20 % of these children will have persistent symptoms with excessive tear secretion, drooling and social problems due to asymmetry in the face. Studies on cortisone treatment to adult patients with acute facial nerve palsy have shown beneficial effects, but no studies with strong quality have been performed in children.

Investigators will perform a double-blind randomized placebo-controlled multicenter trial on children with acute facial nerve palsy. Participants will be recruited consecutively at 9-12 study centers in Sweden during 2019-2020. Oral cortisone (prednisolone) 1 mg/kg x 1 in 10 days (or placebo) will be started on admission. Clinical data, including recovery will be followed-up until 12 months.

The primary outcome is defined as total recovery of the facial nerve palsy, measured with the House-Brackmann scale (grade 1) at 12-months follow-up.

The overall purpose is to assess the utility of cortisone treatment given to children with acute facial nerve palsy in this study. If the total recovery rate is significantly improved in the prednisolone group as compared to the placebo group, prednisolone treatment will be introduced in clinical practice for children with acute facial nerve palsy in order to reduce the risk of persistent symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 1-17 years of age
2. Acute peripheral unilateral facial nerve palsy
3. Less than 72 hours since debut of symptoms
4. Signed informed consent

Exclusion Criteria:

1. Head trauma <1 month
2. Central or bilateral facial nerve palsy
3. Malformations in head and neck
4. Conditions not compatible with cortisone treatment (arterial hypertension, diabetes mellitus, psychiatric disorder, active or latent tuberculosis, intolerance of lactose)
5. Current or past oncological diagnosis
6. Other serious medical conditions (meningitis, encephalitis, stroke)
7. Acute otitis media
8. Signs of herpes simplex or varicella zoster infection (vesicles in the ear region)
9. Pregnancy or breastfeeding
10. Use of any systemic or inhaled steroids within 2 weeks prior onset of symptoms
11. Immunization with live vaccine 1 month prior onset of symptoms
12. Requirement of live vaccine within 2 months from start of experimental treatment (prednisolone or placebo)
13. Evaluation of primary endpoint at 12 months not feasible for any reason
14. Previously included into the FACE study

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
House-Brackmann scale | At 12 months (+/- 2 weeks) after inclusion
  Total recovery in the two treatment groups measured with the House-Brackmann scale.
  The House-Brackmann scale (I is normal function and VI is total loss of function) is chosen as primary outcome measure since it is an objective instrument, easy to perform and the one most frequently used in previous studies. The time point 12 months for evaluation of total recovery is chosen as no further improvement of the facial nerve function is expected after 12 months.

SECONDARY OUTCOMES:
Sunnybrook facial grading system | At 12 months (+/- 2 weeks) after inclusion
  Total recovery in the two treatment groups measured with the Sunnybrook scale.
  The Sunnybrook scale (100 is normal function and 0 is total loss of function) is another objective scale for grading the facial nerve function. It will be used as secondary outcome measure. It is easy to perform and has been used in previous studies in children. It correlates well to the House-Brackmann scale.
Facial Disability Index (FDI) | At 12 months (+/- 2 weeks) after inclusion
  Disease-specific Quality-of-Life assessment scale, with 5 functional domains (5 means no probelms and 2 or 1 means problems all the time) and 5 social domains (6 means problems all the time and 1 means no problems at all)
Facial Clinimetric Evaluation (FaCE) Scale | At 12 months (+/- 2 weeks) after inclusion
  Disease-specific Quality-of-Life assessment scale, with 15 functional and social domains (1 means problems all the time and 5 means no problems at all).
Synkinesis Assessment Questionnaire (SAQ) | At 12 month (+/- 2 weeks) after inclusion
  Subjective grading of synkinesis symptoms with 9 functional domains (1 means no problems at all and 5 means problems all the time).

OTHER OUTCOMES:
Adverse events | Up to 12 month (+/- 2 weeks) after inclusion
  Number of Adverse Events possibly or probably related to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Barbro Hedin Skogman, MD, PhD, Study Director — Center for Clinical Research Dalarna
Locations (15):
- Sweden (15):
  - Barn- och ungdomsmedicin, Falun, Dalarna County
  - Barn och ungdomskliniken, Länssjukhuset, Kalmar, Region Kalmar
  - Barnkliniken, Skaraborgs sjukhus, Skövde, Västra Götalands Region
  - Barnmedicin Drottning Silvias Barn- och Ungdomssjukhus Östra Sjukhuset, Gothenburg
  - Barn- och ungdomsmedicinska kliniken, Jönköping
  - Barn- och ungdomsmottagning, Karlskrona
  - HKH Kronprinsessan Viktorias Barn- och ungdomssjukhus, Linköping
  - Akutmottagning för barn, Skåne Universitets sjukhus, Lund
  - Barnakuten i Malmö, Skåne Universitets sjukhus, Malmo
  - Barn- och ungdomskliniken, Vrinnevi sjukhuset, Norrköping
  - Barn- och ungdomskliniken, Universitets sjukhuset Örebro, Örebro
  - Astrid Lindgrens barnsjukhus, Karolinska Solna, Solna
  - Sachsska barnsjukhuset, Stockholm
  - Astrid Lindgrens barnsjukhus, Karolinska Huddinge, Stockholm
  - Akademisk Barnsjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karlsson S, Arnason S, Hadziosmanovic N, Laestadius A, Hultcrantz M, Marsk E, Skogman BH. The facial nerve palsy and cortisone evaluation (FACE) study in children: protocol for a randomized, placebo-controlled, multicenter trial, in a Borrelia burgdorferi endemic area. BMC Pediatr. 2021 May 4;21(1):220. doi: 10.1186/s12887-021-02571-w. PMID 33947355

DOCUMENTS (2):
  • Study Protocol (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT03781700/Prot_001.pdf
  • Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT03781700/SAP_002.pdf